CLINICAL TRIAL: NCT07162649
Title: A Multicenter, Randomized, Controlled Clinical Trial to Evaluate the Efficacy and Safety of Dexmedetomidine Nasal Spray for the Treatment of Panic Attacks in Adults
Brief Title: Dexmedetomidine Nasal Spray for the Treatment of Panic Attacks in Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yuan Shen (Other)
Collaborators: Shanghai 10th People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Yuan Shen, MD., Ph.D., Tongji University
Organization: Tongji University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: dsyy001
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Experimental): 30μl
  Interventions: Drug: Dexmedetomidine
- Placebo (Placebo Comparator): 30μl
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — 30μl
  Arms: Dexmedetomidine
Drug: Placebo — 30μl
  Arms: Placebo

SUMMARY:
Panic attacks affect 13.2% of adults globally, with acute treatments (e.g., benzodiazepines) carrying dependency risks. Dexmedetomidine, an α₂-adrenergic agonist, achieves peak plasma levels in 5-15 min via nasal delivery and may offer rapid, non-invasive relief for acute panic attacks. Despite preclinical evidence of anxiolytic effects, no randomized trials have evaluated its efficacy for panic attacks.

DETAILED DESCRIPTION:
Panic attacks affect 13.2% of adults globally, with acute treatments (e.g., benzodiazepines) carrying dependency risks. Dexmedetomidine, an α₂-adrenergic agonist, achieves peak plasma levels in 5-15 min via nasal delivery and may offer rapid, non-invasive relief for acute panic attacks. Despite preclinical evidence of anxiolytic effects, no randomized trials have evaluated its efficacy for panic attacks.

This randomized, double-blind, placebo-controlled trial will enroll 400 adults (18-65 years) with DSM-5-defined panic attacks from emergency/outpatient settings. Participants will be randomized 1:1 to dexmedetomidine (30 μg) or placebo nasal spray. The primary outcome is the 30-min response rate (defined as CGI-Efficacy Index >1.0). Secondary outcomes include reduction in core symptom count, anxiety severity (VAS-A), and safety assessments (vital signs, ECG, adverse events). Outcomes will be assessed at baseline, 30 min post-dose, and via telephone follow-ups on Days 7 and 14.

This first RCT of nasal dexmedetomidine for acute panic attacks addresses a critical gap in rapid and non-addictive interventions. It could offer a novel therapeutic option for panic attack patients refractory to first-line treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent is provided after full explanation of objectives, procedures, potential benefits, and risks, with agreement to comply with study requirements.
2. Age between 18 and 65 years at screening.
3. Meet the DSM-5 diagnostic criteria for panic attacks (PA), including but not limited to those occurring in the context of post-traumatic stress disorder, acute stress disorder, generalized anxiety disorder, or social anxiety disorder. At baseline, a Clinical Global Impression-Severity of Illness (CGI-SI) score ≥ 4 is required.
4. Experience an average of ≥2 panic attacks daily during the week preceding enrollment.

Exclusion Criteria:

1. History of panic attacks induced by other psychoactive substances; or prior history of substance abuse involving psychiatric or anesthetic drugs.
2. Use of benzodiazepines, 5-HT1A receptor agonists, or other anxiolytics within 4 hours before enrollment.
3. General anesthesia within the past 28 days.
4. Known hypersensitivity to dexmedetomidine or any component of the investigational product.
5. Myocardial infarction or unstable angina within 6 months; heart rate <60 bpm at screening; history of severe arrhythmias (e.g., Type II second-degree or higher atrioventricular block) or cardiac insufficiency.
6. History of ischemic stroke or transient ischemic attack; uncontrolled hypertension (SBP ≥ 180 mmHg and/or DBP ≥ 110 mmHg) or hypotension (SBP < 90 mmHg and/or DBP ≤ 50 mmHg) despite treatment.
7. Coagulation abnormalities: PT > ULN + 3 s and/or APTT > ULN + 10 s.
8. Significant airway obstruction (e.g., obstructive sleep apnea syndrome, asthma); or use of α2-adrenergic receptor agonists/antagonists within 14 days.
9. Abnormal liver function (ALT/AST >2×ULN or total bilirubin >1.5×ULN) or renal dysfunction (serum creatinine >1.5×ULN).
10. History of cognitive impairment or epilepsy.
11. Pregnant or breastfeeding; or women of childbearing potential unwilling/unable to use effective contraception from 30 days before screening through 6 months after study completion.
12. Any other condition deemed unsuitable by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
30-minute response rate using Clinical Global Impression-Efficacy Index (CGI-EI) | 30 minutes post-administration
  Proportion of participants achieving a CGI-Efficacy Index >1.0 at 30 minutes post-dose, indicating clinically significant symptom improvement. CGI-EI is a validated clinician-rated scale assessing therapeutic effect relative to side effects.

SECONDARY OUTCOMES:
Change in core panic symptom count | Baseline and 30 minutes post-administration
  Reduction in the number of DSM-5-defined core panic symptoms (e.g., palpitations, trembling, choking sensations) self-reported by participants at 30 minutes post-dose.
Change in Visual Analogue Scale for Anxiety (VAS-A) score | Baseline and 30 minutes post-administration
  Reduction in self-reported anxiety severity measured on a 0-10 VAS-A scale (0=no anxiety; 10=maximum anxiety) at 30 minutes post-dose.

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) | 12 hours post-administration
  Frequency of adverse events (e.g., bradycardia, hypotension, nasal irritation, somnolence), serious adverse events (SAEs), abnormal vital signs (BP, HR, RR, SpO₂), and clinically significant ECG changes within 12 hours post-dose.

IPD SHARING:
Plan to Share IPD: No